CLINICAL TRIAL: NCT03909776
Title: A Retrospective Study of Extremity Osteosarcoma Patients Who Recieved Intra-arterial Limb Infusion of Cisplatin During Neoadjuvant Chemotherapy
Brief Title: Transcatheter Intra-arterial Limb Infusion of Cisplatin for Extremity Osteosarcoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBTRA-03/PKUPH-sarcoma 06
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Event-free Survival; Overall Survival; Local-recurrence Free Survival; Pathological Response
Keywords: osteosarcoma; Intra-arterial chemotherapy; survival; Tumor neovascularity; telangiectatic subtype; complications
MeSH Terms: conditions — Osteosarcoma | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IA group (Active Comparator): Cisplatin was given via insertion of a catheter percutaneously by using the Seldinger technique through the brachial or femoral artery under anesthesia and usually at 120 mg/m2 as a 3-h/6-h continuous infusion.
  Interventions: Drug: Cisplatin
- IV group (Sham Comparator): Cisplatin was given at 100-120 mg/m2 as 6-h infusions.
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Cisplatin — Cisplatin was administered intravenously or intraarterially after adequate IV hydration. For IA infusion, cisplatin was given via insertion of a catheter percutaneously by using the Seldinger technique through the brachial or femoral artery under anesthesia and usually at 120 mg/m2 as a 3-h/6-h continuous infusion; while for IV administration, it was given at 100-120 mg/m2 as 6-h infusions.

SUMMARY:
Although there seems to be no benefit from improving the histologic response rate or long-term survival of intra-arterial infusion of cisplatin for localized osteosarcoma of extremities with IOR/OS-3, IOR/OS-5, and COSS 86 protocols, such a treatment strategy is still believed to potentially increase the tumoricidal effect with an increase in higher local concentrations of the infused agents combined with longer tissue exposure time. Besides, the relationship of chemotherapy-induced necrosis and surgical margins is still the main concern for localized osteosarcoma patients to achieve long-term survival. The investigators intend to analyze the gain and loss from transcatheter intra-arterial limb infusion of cisplatin for extremity osteosarcoma in the past six years.

DETAILED DESCRIPTION:
Between December 2009 and August 2014, 119 consecutive extremity osteosarcoma patients were initially treated in Peking University People's Hospital, which were reviewed by the investigators.

The investigators generally recommended neoadjuvant therapy followed by delayed definitive surgery and adjuvant chemotherapy after diagnosis of high-grade osteosarcoma. Patients routinely received neoadjuvant chemotherapy according to the Peking University People's Hospital-Osteosarcoma (PKUPH-OS) regimen, which began in 2008. Generally speaking,the investigators divided neoadjuvant chemotherapy protocols with IA infusion of cisplatin into three small cohorts, and all of these protocols consisted of adriamycin/doxorubicin, cisplatin, and high-dose methotrexate with or without ifosfamide with a time interval of 6-9 weeks. Doxorubicin was usually given for two courses preoperatively, and each course was given as a 3-h pump drip of 2 x 30 mg/m2/d on consecutive days (weeks 0, 6) after cisplatin infusions (weeks 0, 6), followed by two courses of high-dose methotrexate at 8-12 g/m2 with leucovorin rescue, 12 x 9 mg/m2/ i.m. per course. Ifosfamide at 5 x 2.4 g/m2 as 2-h infusions and uromitexan uroprotection was occasionally added to the protocol due to a slow response or huge tumor volume. Cisplatin was administered intravenously or intraarterially after adequate IV hydration. For IA infusion, cisplatin was given via insertion of a catheter percutaneously by using the Seldinger technique through the brachial or femoral artery under anesthesia and usually at 120 mg/m2 as a 3-h/6-h continuous infusion; while for IV administration, it was given at 100-120 mg/m2 as 6-h infusions.

Arteriograms were obtained before the administration of each dose of cisplatin. The last anteroposterior and lateral images obtained in the arteriographic sequence, which demonstrated complete contrast agent filling of the target trunk vessel (i.e., the last full column), were chosen from each arteriogram used for interpretation and comparison with future studies. Only those cases with at least two IA infusions of cisplatin could evaluate the TNV change in tumors. The volume and intensity of TNV on the baseline arteriogram were assessed and compared with those on subsequent arteriograms to assess the rate of change of TNV as an indicator of the tumor response, and only those with more than 90% disappearance of TNV were considered a good response for TNV, or else they were considered a poor response for TNV.

Definitive surgery was scheduled at least 2 weeks after the end of routine cisplatin infusion with the intention of achieving wide surgical margins. All pathology slides were reviewed by two senior pathologists (SKK and SDH). They evaluated all surgical specimens and were blinded to the clinical status. Upon histopathological examination, the tumor response was assessed on the basis of the presence and extent of necrosis, which was determined by a combination of gross and microscopic observations. Tumor necrosis was graded as per Picci et al.[26] histopathological response grading system (Huvos classification), where at least 90% necrosis was defined as a good response and less than 90% necrosis was defined as a poor response. Adjuvant chemotherapy was sequentially performed with the PKUPH-OS protocol for at least 30 weeks after surgery.

Baseline chest CT, bone scans, or positron emission tomography (PET)/CT was used to assess metastatic disease. Patients' follow-up included chest CT, local radiographs, and ultrasound/local CT scans every 3 months, as well as bone scans or PET/CT every 6 months during treatment and two years after completion of adjuvant therapy. During the third to fifth year, chest and pelvic CTs were obtained every 6 months and then yearly thereafter.

Descriptive statistics were used to display demographic data. Kaplan-Meier analysis was used to determine OS, event-free survival (EFS), and recurrence-free survival. The investigators calculated the tumor response rates in different groups as the percentage of patients who had a tumor necrosis rate of more than 90%. The investigators calculated EFS from the date of diagnosis to the last follow-up, local recurrence, distant metastasis, or death. The investigators defined recurrence-free survival from the time of surgery to the date of local recurrence. The investigators compared all the clinical pathological characteristics by Cox univariate analysis of EFS and OS. The investigators also performed subsequent Cox proportional hazards analysis of variables to identify factors associated with survival. Correlation was made between TNV decrease of at least 90% by arteriography and at least 90% tumor necrosis by histologic examination. A P value < 0.05 was considered significant. Analysis was performed using SPSS software package (SPSS Inc., Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* histological diagnosis of high-grade osteosarcoma
* located at extremities
* following the PKUPH-OS protocol
* accept to recieve IA or IV infusion of cisplatin

Exclusion Criteria:

* lost to follow-up
* did not recieve definitve surgery in Musculoskeletal Tumor Center of Peking University People's Hospital
* quiting to recieve chemotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
event-free survival, EFS | 5 years
  We calculated EFS from the date of diagnosis to the last follow-up, local recurrence, distant metastasis, or death.
overall survival, OS | 5 years
  We calculated OS from the date of diagnosis to the last follow-up or death.

SECONDARY OUTCOMES:
pathological response | 2 years
  We calculated the tumor response rates in different groups as the percentage of patients who had a tumor necrosis rate of more than 90%.
recurrence-free survival | 5 years
  We defined recurrence-free survival from the time of surgery to the date of local recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, M.D. and Ph.D., Principal Investigator — Musculoskeletal Tumor Center of Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Xie L, Xu J, Dong S, Gao J, Tang X, Yan T, Yang R, Guo W. Gain and loss from transcatheter intra-arterial limb infusion of cisplatin for extremity osteosarcoma: a retrospective study of 99 cases in the past six years. Cancer Manag Res. 2019 Jul 30;11:7183-7195. doi: 10.2147/CMAR.S214604. eCollection 2019. PMID 31447583